CLINICAL TRIAL: NCT05152095
Title: Therapeutic Effect of Self-administered Auricular Acupressure on Insomnia Induced by Anxiety: A Randomized Sham-controlled Trial
Brief Title: Therapeutic Effect of Self-administered Auricular Acupressure on Insomnia Induced by Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IMU University, Malaysia (Other)
Responsible Party: Principal Investigator, Tang Sin Wei, Lecturer, IMU University, Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCM I-2021 (04)
Record Dates: First submitted 2021-12-01; First posted 2021-12-09 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Insomnia Due to Anxiety and Fear
Keywords: auricular acupressure; insomnia; anxiety; randomized sham controlled trial
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Self-administered Vaccaria seed tapes on auricular acupoints with pressure applied
  Interventions: Other: Vaccaria seed (Wang Bu Liu Xing) pre-attached to adhesive tape used for auricular acupressure
- Sham (Sham Comparator): Self-administered plain tapes (without Vaccaria seed) on auricular acupoints without applying pressure.
  Interventions: Other: Plain ear adhesive tape

INTERVENTIONS:
Other: Vaccaria seed (Wang Bu Liu Xing) pre-attached to adhesive tape used for auricular acupressure — Apply on auricular acupoints, Shenmen and Occiput, apply pressure for 3 minutes, 5 times per day, at the interval of 2 ~ 3 hours, for 5 days.
  Arms: Intervention
Other: Plain ear adhesive tape — Apply on Shenmen and Occiput without applying pressure for 5 days.
  Arms: Sham

SUMMARY:
This is a sham-controlled randomized trial to identify the effectiveness of treating insomnia induced by anxiety with self-administered auricular acupressure in Malaysia.

DETAILED DESCRIPTION:
112 subjects with insomnia and anxiety who fit to the inclusion and exclusion criteria will be recruited into the trial. After initial screening, subjects will be randomly allocated to Vaccaria seed tapes (experimental arm) or non-Varracia seed plain tapes (sham comparator arm).

On the sixth day for the trial (after 5 days of daily auricular acupressure), the ISI and HAM-A score of subjects will be reassessed again. The subjects have to stop applying auricular acupressure for the next five days and reassess their ISI and HAM-A score again on the eleventh day.

ELIGIBILITY:
Inclusion Criteria:

* All Malaysian aged above 18 years old who are suffering from chronic insomnia based on International Classification of Sleep Disorders 3(ICSD-3) and with Insomnia Severity Index (ISI) of 18 and above and more than 3 months.
* Willing to comply with the recommended periodic acupressure stimulation every day during the 1 week period.

Exclusion Criteria:

* Subject with insomnia score below 18 based on Insomnia Severity Index (ISI).
* Subject with stress and anxiety level below 18 in the Hamilton Anxiety Rating Scale (HAM-A).
* Subject with the history of skin sensitivity.
* Subject who just started on new medication to treat insomnia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-11-13 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | 6th day
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Insomnia Severity Index (ISI) | 11th day
  Total score categories:
  0-7 = No clinically significant insomnia 8-14 = Subthreshold insomnia 15-21 = Clinical insomnia (moderate severity) 22-28 = Clinical insomnia (severe)
Hamilton Anxiety Rating Scale (HAM-A) | 6th day
  Total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Hamilton Anxiety Rating Scale (HAM-A) | 11th day
  Total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.

CONTACTS AND LOCATIONS:
Locations (1):
- International Medical University (IMU), Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No